CLINICAL TRIAL: NCT02220192
Title: Focal Loop Electrosurgical Excision Procedure for High-Grade Cervical Intraepithelial Neoplasia: an Alternative Treatment Approach
Brief Title: An Alternative Treatment for Cervical Intraepithelial Neoplasia Using the Focal Loop Electrosurgical Excision Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michelle Khan, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F140613004 (UAB 1425); 000344450-SP012 (Other: Office of Sponsored Programs)
Record Dates: First submitted 2014-08-07; First posted 2014-08-19 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: High-grade Cervical Intraepithelial Neoplasia
Keywords: cervical neoplasia; cervix; high-grade dysplasia; LEEP (loop electrosurgical excision procedure); precancerous cells; colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Focal LEEP (Experimental): All patients will undergo focal treatment of high-grade cervical intraepithelial neoplasia using LEEP. A two-week follow-up assessment will evaluate the side effects of the treatment and any unusual symptoms. This will be done through a phone survey. At six months a clinic visit is required to assess whether there are any precancerous cells of the patient's cervix.
  Interventions: Procedure: Focal LEEP

INTERVENTIONS:
Procedure: Focal LEEP — Focal LEEP may or may not cause less damage to the cervix versus standard LEEP. This could potentially be an advantage by avoiding future complications during pregnancy.

SUMMARY:
This is a pilot study to test the short-term effectiveness of an alternative treatment approach for precancerous cells of the cervix. The study will also explore whether this new treatment is feasible to perform and if it is acceptable to patients.

DETAILED DESCRIPTION:
Standard treatment for precancerous cells of the cervix is called electrosurgical excision procedure (LEEP). Standard LEEP involves treating the entire cervix using FDA-approved equipment. Focal LEEP utilizes the same surgery and the same equipment but only treats the visually unhealthy part of the cervix and not the entire cervix. Side effects and unusual symptoms will be monitored as well as the patient's thoughts and recommendations of the procedure. The total amount of time of study participation is six months.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-45 years old
* Histologically confirmed high-grade cervical intraepithelial neoplasia (CIN2, CIN3, or CIN2/3). A copy of the pathology report is required at the time of enrollment. We will only include patients that had their biopsy performed at the UAB Colposcopy clinic because those that return for treatment represent a select group that is more reliable for follow-up given the standard no-show rate of 50% at the clinic.
* Focal lesion visualized in its entirety colposcopically and involving less than or equal to 2 quadrants of the cervix.
* Satisfactory (adequate) colposcopy.
* Lives within 100 miles of the University of Alabama at Birmingham.

Exclusion Criteria:

* Any suspicion for invasive cancer.
* Glandular abnormalities on cytology or histology.
* Cervical lesion incompletely visualized (e.g. extending into the endocervical canal).
* Endocervical curettage positive for high-grade cervical intraepithelial neoplasia.
* Unreliable for follow-up (drug use, planning to move out of region, etc.). Any patient that lives >100 miles away will be excluded due to concern for possible loss to follow-up.
* Immunosuppression (HIV positive, history of transplantation, lupus on immunosuppressive medication, etc.).
* Pregnancy.
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of cases of recurrent high-grade cervical intraepithelial neoplasia | 6 months
  Recurrence of high-grade cervical intraepithelial neoplasia will be determined from cytologic and/or histologic evidence collected six months following the focal LEEP procedure.

SECONDARY OUTCOMES:
Acceptability of focal LEEP procedure | 2 weeks following focal LEEP procedure
  A 15-minute questionnaire will be conducted by phone with the patient.
Feasibility of focal LEEP of high-grade cervical intraepithelial neoplasia | Within 1 week following focal LEEP procedure
  A short feasibility questionnaire will be completed by the medical provider performing the focal LEEP procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Khan, MD, MPH, Principal Investigator — University of Alabama of Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No